CLINICAL TRIAL: NCT01726751
Title: Spinal Cord Stimulation in the Irritable Bowel Syndrome - a Randomized Cross-over Trial
Brief Title: Spinal Cord Stimulation for Pain Relief in Irritable Bowel Syndrome
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: Medtronics, Inc. (Industry); Bengt Ihre Foundation (Other); The Swedish Society of Medicine (Other)
Responsible Party: Principal Investigator, Per Hellström, Professor, senior consultant, Uppsala University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: SCS-IBS-004
Record Dates: First submitted 2012-10-30; First posted 2012-11-15 (Estimated); Last update posted 2018-11-07 (Actual); Status verified 2018-11

CONDITIONS: Irritable Bowel Syndrome; Constipation; Diarrhea; Pain
Keywords: Spinal cord stimulation; Irritable bowel syndrome; Abdominal pain; Diarrhea
MeSH Terms: conditions — Irritable Bowel Syndrome; Constipation; Diarrhea; Pain; Abdominal Pain

STUDY DESIGN:
Intervention Model Description: Spinal cord stimulation
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early off-stimulation (group B) (Other): Late SCS treatment. After 2 weeks without SCS, randomization to either of two study arms: Group B starting with no SCS for a period of six weeks (A) followed by a period of active SCS (on-period for 6 weeks). Thereafter, free stimulation for 12 weeks, followed by a concluding 2 sweeks of no SCS.
  Interventions: Device: Spinal Cord Stimultion (SCS); Device: Spinal cord nerve stimulation
- Early on-stimulation (group A) (Other): Early SCS treatment. After 2 weeks without SCS, randomization to either of two study arms: Group A starting with SCS for a period of six weeks (A) followed by a period of no SCS (off-period for 6 weeks). Thereafter, free stimulation for 12 weeks, followed by a concluding 2 sweeks of no SCS.
  Interventions: Device: Spinal Cord Stimultion (SCS); Device: Spinal cord nerve stimulation

INTERVENTIONS:
Device: Spinal Cord Stimultion (SCS) — Electric stimulation of the spinal cord
  Other Names: Quad-plus®, Medtronic Inc., MN, USA
Device: Spinal cord nerve stimulation

SUMMARY:
To elucidate Spinal Cord Stimulation (SCS) as treatment for IBS. An SCS system with a 4-polar electrode at the T5-8 level is implanted. In a randomized, cross-over study design, active stimulation is compared to a period without stimulation, with an ensuing tailing stimulation period, twice as long. Patients recorded average pain level, pain attacks, number of diarrheas and global quality of life. At the end of the study patients can choose to retain their SCS stimulation system or have it removed.

The outcome of the present trial will show whether SCS is a useful treatment of IBS. The long-term follow-up will show the continuous amelioration of SCS over at least six months.

DETAILED DESCRIPTION:
The primary aim of the study is to investigate if the typical chronic abdominal pain in IBS can be ameliorated by SCS. Secondary aims are possible effects of SCS on diarrhea or constipation, quality of life and side effects, and further to evaluate the feasibility and tolerability of SCS as validated by the willingness of the patients to retain the SCS stimulation equipment.

Eligible patients are selected by a gastroenterologist for the study inclusion criteria: age 18-60, fulfilment of Rome II criteria, abdominal pain episodically reaching > 4 on a 0-10 VAS, and stable symptoms for the past 2 years. A thorough clinical work-up is done to exclude organic disease, including routine blood and electrolyte status, hepatic enzyme function and lactose tolerance test as well as colonoscopy or colon x-ray. Patients with significant somatic or psychiatric co-morbidity will be excluded.

Study design: A quadripolar SCS-lead (Quad-plus®, Medtronic Inc., Minnesota, USA) was implanted via a percutaneous puncture at the Th11/12 level of the dorsal epidural space in local anesthesia with the patient in the prone position. The electrode is advanced to the mid-thoracic level, aiming for a final position around T6-T8, until intraoperative stimulation yields paresthesias covering the abdomen . The electrode is then connected to an impulse generator (Itrel-3®, Medtronic Inc.) implanted subcutaneously in the upper left quadrant of the abdomen. Stimulation frequency will be set to 50 Hz for all patients but other parameters (electrode pole combinations, amplitudes and pulse width) are adjusted and set to produce adequate paresthesias of comfortable intensity.

During the subsequent ongoing trial reprogramming was allowed, if necessary for optimal stimulation.

SCS will be started 2 weeks after surgery. Thereafter patients are randomized to either of two study arms: one starting with SCS for a period of six weeks (A), and another with six weeks without SCS (delayed start) (B). When on active SCS, patients are prompted to stimulate 8-12 h per day. Patients are instructed to increase the stimulation upon pain attack break-through.

After six weeks, patients without stimulation were crossed-over to stimulation and vice versa. After another six weeks both study arms included continued stimulation for additional 12 weeks up to 26 weeks. After a final 2-week period without stimulation the trial is terminated.

During the whole study period patients will record, on a daily basis: 1) number of pain attacks, 2) number of diarrhea episodes, 3) average pain level for the day (0-10) and 4) average quality of life (0-10).

Patients are scheduled for regular controls, at 2, 8, 14, 26 and 28 weeks after implantation. Patient compliance will be ensured, as the impulse generator stores information on the percentage of elapsed time that stimulation has been in use.

At termination of the study participants were offered to keep the implanted SCS system or have it removed.

All patients will be contacted for a structured telephone interview follow-up at a time-point varying between 18 to 78 months after the study termination. A questionnaire was used to assess present pain level, medication, use of the SCS system, side effects and global satisfaction. Patients will also be asked whether they would have participated if they had known the outcome in advance, and if they would recommend a trial of SCS treatment to someone else with similar gastrointestinal problems.

All patients will be evaluated with the hospital anxiety and depression scale (HADS) and a modified version of the gastrointestinal symptom rating scale for IBS (GSRS-IBS).

ELIGIBILITY:
Inclusion Criteria:

* age 18-60, Rome II criteria, abdominal pain >4 (0-10 VAS), stable symptoms for >2 years

Exclusion Criteria:

* other gastrointestinal disease, somatic or psychiatric co-morbidity

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2005-08; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
To investigate if typical abdominal pain of IBS can be ameliorated by SCS? | According to protocol for 26 weeks
  During the whole study period each patient will record the number of pain attacks.
  Patients are scheduled for regular outpatient controls, at 2, 8, 14, 26 and 28 weeks after implantation

SECONDARY OUTCOMES:
To record effects of SCS on diarrhea/constipation | According to protocol for 26 weeks
  During the whole study period each patient recorded, on a daily basis: 1) number of pain attacks, 2) number of diarrhea episodes, 3) average pain level for the day and 4) assessment of average quality of life. For the latter two items patients were instructed to use a numerical rating scale (NRS) with a range of 0-10.
  Patients were scheduled for regular outpatient controls, at 2, 8, 14, 26 and 28 weeks after implantation

OTHER OUTCOMES:
To evaluate quality of life and side effects, feasibility and tolerability of SCS, validated as willingness to retain the stimulation equipment. | According to protocol for 26 weeks
  During the whole study period each patient recorded, on a daily basis: 1) number of pain attacks, 2) number of diarrhea episodes, 3) average pain level for the day and 4) assessment of average quality of life. For the latter two items patients were instructed to use a numerical rating scale (NRS) with a range of 0-10.
  Patients were scheduled for regular outpatient controls, at 2, 8, 14, 26 and 28 weeks after implantation.

CONTACTS AND LOCATIONS:
Overall Officials: Per M Hellström, MD, PhD, Principal Investigator — Uppsala University
Locations (1):
- Karolinska University Hospital, Solna, Stockholm County, Sweden

REFERENCES:
- [Derived] O'Connell NE, Ferraro MC, Gibson W, Rice AS, Vase L, Coyle D, Eccleston C. Implanted spinal neuromodulation interventions for chronic pain in adults. Cochrane Database Syst Rev. 2021 Dec 2;12(12):CD013756. doi: 10.1002/14651858.CD013756.pub2. PMID 34854473